CLINICAL TRIAL: NCT03129464
Title: Effect of Cold Therapy Implementation on Multi-modal Postoperative Pain Management in Women Undergoing Laparoscopic Hysterectomy
Brief Title: Effect of Cold Therapy Implementation on Multi-modal Postoperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, Pamela Frazzini Padilla, Clinical Fellow, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FLA 16-111
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cold Therapy (Experimental): Patients undergoing total laparoscopic hysterectomy will receive routine pre-operative multi-modal analgesia regimen and well as routine post-operative analgesia with instructions for dosing. Intervention will include the patient being asked to use a reusable cold gel pack to deliver cold therapy to their abdominal incisions every 6 hours for the first 72 hours.
  Interventions: Device: Cold therapy via reusable cold gel pack
- Control (No Intervention): Patients undergoing total laparoscopic hysterectomy will receive routine pre-operative multi-modal analgesia regimen and well as routine post-operative analgesia with instructions for dosing. They will not receive any additional intervention.

INTERVENTIONS:
Device: Cold therapy via reusable cold gel pack — Patients in the experimental group will be asked to apply cold therapy to their abdominal incisions every 6 hours for the first 72 hours following their surgery (total laparoscopic hysterectomy). Cold therapy will be applied via a reusable cold gel pack.
  Arms: Cold Therapy

SUMMARY:
This is a pilot randomized controlled trial examining post-operative pain scores and outcomes after laparoscopic hysterectomy in patients prescribed cold therapy as an adjunct to routine post-operative multi-modal analgesia, compared to those patients prescribed routine multi-modal analgesia without cold therapy. All patients scheduled for total laparoscopic hysterectomy (without robotic-assistance) will be screened for eligibility in the study. If eligible, patients will be invited to participate in the study and standardized informed consent process will ensue. After surgery is completed participants will be randomized to either the control group or the study group. The study group will be prescribed the use of cold therapy to their abdominal incisions through reusable cold gel packs. The cold therapy is to be applied to participants' incisions for the first three postoperative days, in addition to routine post-operative analgesia regimen. Investigators will then collect information on pain scores, narcotic use, quality of life and surgical recovery scores.

This study aims to examine if there is a difference in post-operative pain scores with the application of cold therapy to laparoscopic abdominal incisions following laparoscopic hysterectomy, when compared to no cold therapy. Secondarily, investigators will examine post-operative quality of life scores, postoperative surgical recovery scores, as well as narcotic use among the two groups. Investigators also aim to ascertain additional information regarding total quantity of narcotics used post-operatively to aid in prescribing patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Patients can understand and voluntarily sign an informed consent form
2. Female gender ages 18-65
3. Scheduled for laparoscopic hysterectomy for benign indications, total or subtotal, without or without oophorectomy (standard of care involves bilateral salpingectomy)

Exclusion Criteria:

1. Conversion to laparotomy
2. Diagnosis of chronic pelvic pain
3. No access to freezer at home to keep reusable cold packs cold between uses
4. Contraindications to exposure to cold therapy (history of cold allergy, cold intolerance, Raynaud's disease, cold urticaria, cryoglobulinemia, or pyoderma gangrenosum)
5. Medical contraindication to NSAID use

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Sprague, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Therapy | Control
Started | 28 | 28
Completed | 28 | 27
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Therapy | Control | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (5.8) | 47.2 (6.19) | 46.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 8 | 12 | 20
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Score
Description: Post-operative pain score on an 11 point numeric rating scale, minimum value of 0 and maximum value of 10, zero meaning no pain and 10 meaning the worst pain imaginable.
Time Frame: 24 hours post-operatively following total laparoscopic hysterectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 28 | 27
units on a scale | 4 [2 to 6] | 4.5 [3 to 5.75]

2. Secondary Outcome: Post-operative Pain Score
Description: as for outcome 1
Time Frame: 72 hours post-operatively following total laparoscopic hysterectomy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 25 | 27
score on a scale | 2 [1 to 4] | 2.5 [1.25 to 5.75]

3. Secondary Outcome: Patient Reported Quantity of Narcotics Used Post-operatively
Description: Patient reported quantity of narcotics used post-operatively measured in number of reported 5 mg oxycodone tabs consumed
Time Frame: 72 hours post-operatively following total laparoscopic hysterectomy
Measure: Mean (Standard Deviation); unit: oxycodone tabs
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 25 | 27
oxycodone tabs | 2.52 (2.97) | 4.78 (6.32)

4. Secondary Outcome: Quality of Life Score as Measured by the Validated Abdominal Surgery Impact Scale
Description: Quality of life score as measured by the validated Abdominal Surgery Impact Scale, minimum value is 18, maximum value is 126, with lower values indicating a worse quality of life and higher scores indicating a better quality of life.
Time Frame: 72 hours post-operatively following total laparoscopic hysterectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 25 | 27
score on a scale | 43.8 (11) | 45.7 (18)

5. Secondary Outcome: Surgical Recovery Score as Measured by the Validated Surgical Recovery Scale
Description: Functional surgical recovery following major surgery as measured by the validated Surgical Recovery Scale, possible scores range from 0 to 60, with higher scores indicating a better recovery
Time Frame: 10-14 days post-operatively following total laparoscopic hysterectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 28 | 28
score on a scale | 39.7 (9.68) | 38 (10.1)

6. Other Pre Specified Outcome: Total Amount of Narcotics Used Post-operatively
Description: Total amount of narcotics used post-operatively within the first two weeks after surgery measured in MME, intravenous morphine milligram equivalents.
Time Frame: 10-14 days postoperatively following total laparoscopic hysterectomy
Measure: Mean (Standard Deviation); unit: MME, intravenous morphine milligram equi
Arm/Group | Cold Therapy | Control
Number analyzed (Participants) | 28 | 28
MME, intravenous morphine milligram equi | 13.3 (12) | 23.7 (23.6)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Cold Therapy | Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT03129464/Prot_SAP_000.pdf